CLINICAL TRIAL: NCT00918450
Title: A Phase 2b Monotherapy Study of ABT-263 in Subjects With Relapsed or Refractory B-Cell Chronic Lymphocytic Leukemia
Brief Title: Study Assessing the Safety and Efficacy of ABT-263 in Subjects With B-cell Chronic Lymphocytic Leukemia (CLL) Who Have Failed at Least One Prior Fludarabine-containing Regimen
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor has decided to not proceed with this study.
Sponsor: Abbott (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sari Enschede, MD, Abbott Laboratories
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M10-738
Record Dates: First submitted 2009-05-22; First posted 2009-06-11 (Estimated); Last update posted 2010-02-26 (Estimated); Status verified 2010-02

CONDITIONS: B-cell Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — navitoclax

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ABT-263

INTERVENTIONS:
Drug: ABT-263 — Continuous dosing until disease progression using one of the following formulations:
  25 mg/mL oral solution OR 50 mg/mL oral solution OR 2.0 grams/bottle powder for oral solution of 25 mg/mL when mixed OR 2.0 grams/bottle powder for oral solution of 50 mg/mL when mixed

SUMMARY:
This is a Phase 2b, open-label, multicenter, global study assessing the safety and efficacy of ABT-263 in subjects with B-cell CLL who have failed at least one prior fludarabine-containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 yrs of age, have B-cell CLL, failed at least 1 prior fludarabine-containing regimen.
* Refractory to 1 fludarabine-containing regimen is defined as failure to achieve at least PR to the last fludarabine-containing regimen received, or disease progression while receiving the last fludarabine-containing regimen, or disease progression in responders (i.e., achieved a PR or CR) within 6 mos of the last cycle of the last fludarabine-containing regimen received (e.g., fludarabine monotherapy, FR, or FC) or in responders (i.e., achieved a PR or CR ) within 24 mos of the last cycle of FCR.
* Intolerant to fludarabine is defined as discontinuation of therapy within 2 cycles due to side effects/toxicity from the last fludarabine-containing regimen.
* ECOG score of <=1.
* Adequate coagulation, renal, & hepatic function at Screening as follows:

  * Serum creatinine <= 2.0 mg/dL or calculated creatinine clearance >= 50 mL/min;
  * AST & ALT <= 3.0 x ULN;
  * Bilirubin <= 1.5 x ULN.
* Gilbert's Syndrome may have a Bilirubin > 1.5 x ULN; aPTT, PT, not to exceed 1.2 x ULN.
* Adequate bone marrow (BM) independent of any growth factor support (with the exception of subjects with BM heavily infiltrated with underlying disease [80% or more] who may use growth factor support to achieve adequate BM) at Screening as follows:

  * ANC >= 1000/µL;
  * Platelets >= 75,000/mm3 (entry platelet count must be independent of transfusion within 14 days of Screening);
  * Hemoglobin >= 9.0 g/dL.
* History of autologous BM transplant must be > 6 mos post transplant (prior to the 1st dose of study drug) & have adequate BM independent of any growth factor support (with the exception of subjects with BM that is heavily infiltrated with underlying disease [80% or more] who may use growth factor support to achieve adequate BM) at Screening as follows:

  * ANC >= 1500/µL;
  * Platelets >= 125,000/mm3;
  * Hemoglobin >= 10.0 g/dL.
* Female subjects must be surgically sterile, postmenopausal (at least 1 year), or have negative results on a pregnancy test.
* All female subjects not surgically sterile or postmenopausal (at least 1 year) & non-vasectomized male subjects must practice birth control.

Exclusion Criteria:

* History/clinically suspicious for cancer-related CNS disease.
* Undergone allogeneic stem cell transplant.
* Undergone autologous stem cell transplant w/i 6 mos prior to 1st dose.
* History/predisposing condition of bleeding or currently exhibits signs of bleeding.
* Recent history of non-chemotherapy induced thrombocytopenic associated bleeding w/i 6 mos prior to 1st dose.
* Active peptic ulcer disease or other hemorrhagic esophagitis/gastritis.
* Active immune thrombocytopenic purpura or history of being refractory to platelet transfusions w/i 1 yr prior to 1st dose.
* Currently receiving/requires anticoagulation therapy or any drugs or herbal supplements that affect platelet function, with the exception of low-dose anticoagulation medications used to maintain the patency of a central IV catheter.
* Significant history of cardiovascular disease, renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, or hepatic disease.
* Positive for HIV, Hepatitis B, or Hepatitis C.
* Previous or current malignancies w/i the last 3 yrs:

  * except adequately treated in situ carcinoma of the cervix uteri;
  * basal or squamous cell carcinoma;
  * in situ carcinoma of the bladder;
  * or previous malignancy confined and surgically resected with curative intent.
* Has Prolymphocytic leukemia or Richter's transformation to an aggressive B-cell malignancy.
* Exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to uncontrolled systemic infection or diagnosis of fever and neutropenia w/i 1 week prior to study drug.
* Prior exposure to ABT-263.
* Received antibody therapy w/i 30 days prior to 1st dose.
* Received any anti-cancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal, or any investigational therapy w/i 14 days prior to the 1st dose, or has not recovered to <Gr2 clinically significant AE(s) /toxicity(s) of the previous therapy.
* Received steroid therapy for anti-neoplastic intent, w/i 7 days prior to the 1st dose with the exception of inhaled steroids for asthma, topical steroids, or replacement/stress corticosteroids.
* Received aspirin w/i 7 days prior to the 1st dose.
* Consumed grapefruit or grapefruit products w/i 3 days prior to 1st dose.
* Females pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Assess the safety of ABT-263 by evaluating study drug exposure, adverse events, serious adverse events, all deaths, as well as changes in laboratory determinations and vital sign parameters. | monthly (at a minimum)
Assess the objective response rate (partial response [PR] and confirmed complete response [CR]) of B-cell CLL subjects treated with ABT-263. | Every 3 months

SECONDARY OUTCOMES:
Assess the effects of ABT-263 on duration of overall response, PFS and overall survival in subjects with B-cell CLL. | Every 3 months
Assess the effects of ABT-263 on time to response, 12-month survival rate, time to disease progression (TTP), and disease control rate in subjects with B-cell CLL . | Every 3 months
Investigate the effects of ABT-263 on quality of life (FACT-Leu and EQ-5D), ECOG performance status, and biomarkers in subject with B-cell CLL. | Every 3 months